CLINICAL TRIAL: NCT05540704
Title: Changing the T1DE (Type 1 Disordered Eating): A Randomized Controlled Trial Comparing ACT to Supportive Diabetes Counseling
Brief Title: Study Comparing Acceptance and Commitment Therapy (ACT) to Supportive Diabetes Counseling for Problematic Eating and Weight Control in Type 1 Diabetes
Acronym: T1DE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00111401; 4-SRA-2022-1226-M-B (Other Grant/Funding Number: Breakthrough T1D (formerly JDRF))
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Eating Disorders; Disordered Eating Behaviors; Purging (Eating Disorders); Binge-Eating Disorder
Keywords: T1DE; "diabulimia"; glycemic control; disordered eating behavior; eating disorders; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders; Disordered Eating Behavior; Binge-Eating Disorder; Diabulimia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded to the participant's assignment/condition. All study team members are blinded to the randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy for Type 1 Diabetes - Eating Disorder (ACT-T1DE) (Experimental): ACT-T1DE consists of 12 sessions of flexible ACT protocol tailored to the unique conditions and needs of type 1 diabetes eating disorders. The protocol is based on an initial pilot study (Merwin et al., 2021); however, the current protocol has been modified, based on key stakeholder feedback and to optimize real-world implementation. Modifications include transition from the use of a mobile app to a text messaging platform and a combination of in-person and virtual visits.
  Interventions: Behavioral: iACT
- Supportive Diabetes Counseling (SDC) (Active Comparator): The SDC condition is a flexible protocol of 12 sessions consisting of supportive listening, diabetes-related psychoeducation and goal setting, based on the ADA Type 1 Diabetes Self-Care Manual and ADCES7 Self-Care Behaviors.
  Interventions: Other: Supportive Diabetes Counseling

INTERVENTIONS:
Behavioral: iACT — Treatment is based on Acceptance and Commitment Therapy (ACT), a contemporary cognitive behavioral therapy (CBT) that improves human functioning and adaptability by increasing psychological flexibility. Individual therapy sessions are paired with mobile phone delivered interventions.
  Arms: Acceptance and Commitment Therapy for Type 1 Diabetes - Eating Disorder (ACT-T1DE)
Other: Supportive Diabetes Counseling — 12 sessions of counseling with a diabetes educator knowledgeable about disordered eating in type 1 diabetes. Intervention focuses on supportive listening, diabetes-related education and goal setting.
  Arms: Supportive Diabetes Counseling (SDC)

SUMMARY:
The goal of this study is to test the effectiveness of two different approaches to treating problematic eating and weight control in type 1 diabetes. Participants are between the ages of 16-50 and complete 12 sessions of either Acceptance and Commitment Therapy (ACT) or Supportive Diabetes Counseling over 16 weeks. They use their mobile phone between sessions to increase engagement and reinforce learning.

The main questions are:

Do participants show improvements in glycemic levels, eating disorder symptoms, diabetes management and diabetes distress?

Does one treatment do better than the other?

How do the treatments work, if they work, and for whom?

Participants complete assessments that include wearing a continuous glucose sensor and activity watch, and get a blood draw to determine HbA1c. They also complete diagnostic interviews, surveys and computer tests of attention and reactions. These assessments help us better understand the types of changes that are happening and how they might influence health and well-being.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing Acceptance and Commitment Therapy (ACT) to supportive diabetes counseling (SDC) for individuals with type 1 diabetes (T1D) and disordered eating (or T1DE). Both conditions are tailored to the unique needs of individuals living with T1D and the unique conditions under which an eating disorder develops and is maintained. Participants will be 128 individuals with T1D, between the ages of 16-50, with binge-purge eating disorders (EDs), including threshold and subthreshold bulimia nervosa, binge eating disorder and purging disorder. Purging includes restriction of insulin for weight loss. An expansion cohort of 58 persons with T1D and elevated Diabetes Eating Problems Survey-Revised scores (DEPS-R=>20) will also be recruited to assess the utility of the protocol for a broader array of eating problems in T1D. Participants will be randomized to either ACT or SDC, and complete assessments at baseline, mid-treatment, end-of-treatment, 1 month, 3 months, and 6 months post-treatment. The primary outcome of interest for power and sample size calculation is mean blood glucose as assessed by continuous glucose monitoring. Other outcomes include hemoglobin A1c (HbA1c), eating disorder symptoms, diabetes self-management and, secondary, diabetes distress. In addition to examining clinical outcomes, this study tests biobehavioral mechanisms of change and predictors of treatment response. Process of change assessments focus on flexible responding to pathology-relevant stimuli and early improvement in glycemic control affecting executive function. The primary site is Duke University Medical Center. The Miriam Hospital is a secondary site.

ELIGIBILITY:
Primary Cohort

Inclusion Criteria:

* 16-50 years of age
* Diagnosis of Type 1 diabetes
* Eating disorder characterized by binge eating and/or problematic weight control behaviors, including withholding insulin (Bulimia Nervosa, Binge Eating and Purging Disorder spectrum diagnoses)
* Independently manages diabetes (not reliant on a caregiver)

Expansion Cohort

Inclusion Criteria:

* 16-50 years of age
* Diagnosis of Type 1 diabetes
* DEPR-R score >=20 but does not meet criteria for the primary cohort

Primary and Expansion Cohort

Exclusion Criteria:

* Active suicidal ideation
* Diagnosis of Avoidant Restrictive Food Intake Disorder or Anorexia Nervosa spectrum diagnoses
* Hypoglycemic unawareness as assessed by the Gold Method and multiple severe episodes of hypoglycemia requiring 3rd party assistance in the last 2 years
* Current substance abuse disorder or current or past psychotic disorder
* NonEnglish speaking

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic control as indexed by continuous glucose monitoring (CGM) | baseline, 6 weeks, 12 weeks, 36 weeks
  CGM indices of time in range, frequency of Level 1 and 2 hyperglycemia and blood glucose variability
Change in eating disorder symptoms as indexed by the Diabetes Eating Problems Survey-Revised (DEPS-R) | baseline, 12 weeks, 16 weeks, 24 weeks, 36 weeks
  Severity of eating and body image concerns, frequency of engagement in maladaptive eating and weight control behaviors, specifically in the context of diabetes. Scores range from 0-80, with higher scores indicating greater symptom severity (worse outcome).
Change in diabetes self-management as indexed by the Diabetes Self-Management Questionnaire | baseline, 12 weeks, 16 weeks, 24 weeks, 36 weeks
  Engagement in activities necessary to manage diabetes, including checking blood sugar and administering insulin. Scores range from 0-10 with higher scores indicating better self-management.
Change in glycemic control as indexed by hemoglobin A1c (HbA1c) | baseline, 24 weeks, 36 weeks
  Glycated hemoglobin (percentage of red blood cells that are glycated providing an estimate of average blood glucose over 3 months)

SECONDARY OUTCOMES:
Change in diabetes distress as indexed by the Type 1 - Diabetes Distress Scale | baseline, 12 weeks, 24 weeks, 36 weeks
  Feelings of stress or overwhelm with the burden of living with diabetes and diabetes management. Scores range from 1-6, with higher scores indicating greater distress (worse outcome)
CompACT-10 | Baseline, Mid-Treatment, 12 weeks, 16 weeks, 24 weeks, 36 weeks.
  A 10-item measure of general (rather than diabetes-specific) psychological flexibility. This measure includes component processes of open, aware and engaged, allowing for more in-depth assessment of process of change. This is the primary psychological flexibility measure in the current trial.
Acceptance and Action Diabetes Questionnaire (AADQ) | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Assesses psychological flexibility (process of change) in the context of diabetes specific thoughts and feelings.
Valuing Questionnaire (VQ) | Baseline, 6 weeks, 12 weeks, 24 weeks, 36 weeks
  Assesses outcomes expected in an ACT intervention. The VQ consists of 2 Subscales: Values Obstruction and Values Progress. Values Obstruction measures the extent to which thoughts/feelings obstructed engagement in values. Values Progress measures the extent to which an individual made progress in areas of life that are important to them.
Executive function | Baseline, 12 weeks, 36 weeks
  Computer-administered Stroop and a GoNoGo paradigm. Outcomes of interest are interference or bias score and errors and reaction time (respectively). These measures are included to test the hypothesis that executive function is improved with the improvement of eating disorder symptoms and glycemic control.
High Frequency Heart Rate Variability (HF-HRV) | Baseline, 12 weeks, 36 weeks
  Assesses physiological flexibility/adaptability in the presence of emotional stimuli as an exploratory process of change measure.
Actigraphy | Baseline, 12 weeks, 36 weeks
  Measures sleep and physical activity as exploratory measures of behavioral mechanisms of change.
Ecological Momentary Assessment (EMA) | Baseline, 12 weeks, 36 weeks
  Participants complete questions at home using their mobile phone assessing psychological flexibility, mood, eating and diabetes management behavior, for additional data with high ecological validity. The assessment also aims to test the hypothesis that negative mood is decoupled from problem behavior over the course of treatment.
Change in Eating Disorder Examination - Questionnaire (EDE-Q) | Baseline, 16 weeks, 24 weeks, 36 weeks
  Self-report version of the Eating Disorder Examination (EDE). The EDE includes a total score and 4 subscale scores: Restraint, Eating Concerns, Weight Concerns, Shape Concerns. It is included to capture aspects of ED not assessed by the DEPS, as well as diagnostic outcome or change.
GAD-7 | Baseline, 12 weeks, 36 weeks
  7-Item assessment of anxiety. The primary purpose for inclusion is as a control variable.
PHQ-9 | Baseline, 12 weeks, 36 weeks
  9-Item assessment of Depression. The primary purpose for inclusion is as a control variable.
T1DE Questionnaire | Baseline, End-of-Treatment, 3 Months, 6 Months
  This is a 20-item questionnaire developed for the purposes of this trial. The questionnaire is an inventory of target behaviors for individuals with T1DE.

OTHER OUTCOMES:
Working Alliance Inventory - Short Revised | Mid-treatment
  This is a 13-item self-report questionnaire that measures experiences individuals have with their therapy or therapist. It includes three subscale scores: goal items, task items, and bond items. It is included as a potential moderator of treatment effects.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Merwin, PhD, Principal Investigator — Duke University faculty
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No